CLINICAL TRIAL: NCT06190964
Title: Assessing the Impact of Integrative Medicine on Anxiety and Wellbeing of Hospital Workers Exposed Directly or Indirectly to Terror, Trauma or War
Brief Title: Integrative Medicine for Hospital Workers Exposed to War
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0105-23-BNZ
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Anxiety
Keywords: Acute Stress Disorder; Anxiety; Integrative medicine; Hospital workers; War
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Traumatic, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrative medicine (Experimental): The employees are treated by a team from the system for integrative medicine, including practitioners of acupuncture; touch/movement techniques (for example, qigong, reflexology, shiatsu) or mind-body medicine (for example, relaxation and breathing exercises) and may include one or more of the above 3 treatment areas.
  Interventions: Other: Integrative medicine

INTERVENTIONS:
Other: Integrative medicine — Acupuncture; touch/movement techniques (for example, qigong, reflexology, shiatsu) and/or mind-body medicine (for example, relaxation and breathing exercises)

SUMMARY:
During the "Iron Swords" war in Israel in 2023, the residents of the Gaza Strip and the surrounding area, along with the soldiers of the security service, were exposed to a very high intensity of trauma. Added to this is an extensive cycle of trauma for those who were directly and indirectly exposed to loss and terror throughout the country. Medical teams in the hospitals and in the community were exposed with the highest intensity to these traumatic aspects which were amplified by the collapse of many of the resilience and mental health centers in the south.

An integrative medicine treatment clinic was established at the Bnai Zion Medical Center for the purpose of providing a response to all hospital employees who are exposed and will be exposed (directly or indirectly) to the wounded and patients expressing trauma, including symptoms of acute stress disorder, as a result of war and terrorism. Hospital employees are invited to register for complementary medicine treatments on the hospital's website according to indications that include anxiety, emotional distress and/or typical Acute Stress Disorder (ASD) symptoms, including physical distress (such as pain, breathing disorder, digestive system symptoms, exhaustion, etc.). The employees are treated by a team from the system for integrative medicine, including practitioners of acupuncture; touch/movement techniques (for example, qigong, reflexology, shiatsu) or mind-body medicine (for example, relaxation and breathing exercises) and may include one or more of the above 3 treatment areas.

In the proposed study, the investigators plan to examine the effect of these treatments on various symptoms experienced by hospital employees during this period.

ELIGIBILITY:
Inclusion Criteria:

* Hospital employees
* Anxiety, emotional distress and/or typical ASD symptoms directly or indirectly related to exposure to the trauma of terrorism or war

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-10-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptom relief | Before intervention; 24 hours after intervention
  Measure Yourself Concerns and Wellbeing (MYCAW) questionnaire: minimum value: 0; maximum value: 6; higher score means worse outcome.

SECONDARY OUTCOMES:
Stress and anxiety | Before intervention; 4 to 8 weeks after intervention
  Acute Stress Disorder (ASD) questionnaire: minimum value: 0; maximum value: 63; higher score means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Attias, PhD, Principal Investigator — Complementary Medicine Service
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/64/NCT06190964/Prot_SAP_000.pdf